CLINICAL TRIAL: NCT02892708
Title: Impact of Surgery on the Treatment of Supratentorial Malignant Gliomas in Subjects Aged 70 and Over
Acronym: CSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K060215; ID RCB : 2007-A00522-51 (Other: ANSM)
Record Dates: First submitted 2016-05-17; First posted 2016-09-08 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Malignant Glioma
Keywords: supratentorial gliomas; surgery; magnetic resonance spectroscopy; elderly
MeSH Terms: conditions — Glioma | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Active Comparator): Surgical resection followed by radiation therapy
  Interventions: Procedure: Surgery
- radiotherapy alone (Experimental): radiotherapy after a brain biopsy
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Procedure: Surgery — partial or complete resection followed by radiotherapy
  Arms: Surgery
Radiation: radiotherapy — radiotherapy after a brain biopsy
  Arms: radiotherapy alone

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of surgical resection in elderly patients 70 years or older with a supratentorial glioblastoma de novo. The sensitivity of Magnetic Resonance Spectroscopy with perfusion sequences in the diagnosis of malignant glioma in the elderly will also be studied.

DETAILED DESCRIPTION:
Currently, the standard treatment for gliomas is based on surgical resection followed by radiation therapy.

However in patients 70 and older, surgery is not systematic, before radiotherapy. Moreover, at these ages, surgery is likely to be less well tolerated in general terms.

The aim of this study is to try to determine the best treatment between radiation therapy associated with the surgical treatment and care by radiotherapy alone, after a brain biopsy. This is a randomized, two arms, multicenter, open study.

In the two weeks following the radiological diagnosis of a lesion highly suggestive of a high-grade glioma, patients will be randomized to either arm surgery (partial or complete excision) + radiotherapy or in the radiotherapy alone arm. Within 5 weeks after surgery (biopsy or excision), all patients will receive treatment with focal radiotherapy.

A central review blades and MRI data will be organized after the inclusion of patients.

A maximum of 135 patients will participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Highly suggestive radiological aspect of a high-grade glioma
* Operability of the lesion, defined according to standard criteria of literature: lobar tumor, cortico-subcortical, well limited, without deep infiltration and without involvement of the basal ganglia. This operability is to reassess based on surgical experience and the ability to remove more or less completely a tumor of this type in a given location
* Age greater than or equal to 70 years
* Preoperative Karnofsky Index ≥ 50
* Information given to the patient or his family and signed written consent.

Exclusion Criteria:

* Existence of a cons-indication to MRI
* Non operability of the lesion
* Unbalanced concomitant serious pathology that might be an indication against-formal anesthetic (ASA 4-5) (see annex)
* Previous history of radiotherapy or chemotherapy prior to this injury
* Patient under guardianship or under judicial protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
duration of survival | From date of randomization until the date of death from any cause, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cornu, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Florence Laigle, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laigle-Donadey F, Metellus P, Guyotat J, Menei P, Proust F, Dufour H, Chinot O, Honnorat J, Faillot T, Paquis P, Peruzzi P, Emery E, Guillamo JS, Carpentier A, Wager M, Lebbah S, Hajage D, Delattre JY, Cornu P. Surgery for glioblastomas in the elderly: an Association des Neuro-oncologues d'Expression Francaise (ANOCEF) trial. J Neurosurg. 2022 Oct 14;138(5):1199-1205. doi: 10.3171/2022.8.JNS221068. Print 2023 May 1. PMID 36242578